CLINICAL TRIAL: NCT05341466
Title: Examining the Relationship Between Changes in Corticospinal Excitability and Motor Learning After Acute Intermittent Hypoxia in Able-bodied Individuals for Subsequent Study in Individuals With Incomplete Spinal Cord Injury.
Brief Title: The Effect of Acute Intermittent Hypoxia on Motor Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Colorado, Denver (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Andrew Quesada Tan, Assistant Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-3980; P2CHD086844 (NIH)
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Incomplete Spinal Cord Injury
Keywords: Spinal Cord Injury; Motor Adaptation; Acute Intermittent Hypoxia
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This study design is twofold. The first study examines the effects of AIH on motor learning using an AIH group and a control group (total N = 30). The second part of this study examines corticospinal indices of motor learning using an AIH group and a SHAM group (i.e., blinded normoxia; total N = 26).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Repetitive Acute Intermittent Hypoxia (Experimental): 5 consecutive days of 15, 1.5 min episodes at 9% O2 (AIH) alternating with 21% O2 at 1 min intervals
  Interventions: Other: Acute Intermittent Hypoxia
- SHAM Acute Intermittent Hypoxia (Sham Comparator): 5 consecutive days of 15, 1.5 min episodes at 21% O2 (SHAM AIH) alternating with 21% O2 at 1 min intervals
  Interventions: Other: SHAM Acute Intermittent Hypoxia
- Control (No Intervention): The control group received no AIH exposure.

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — 5 consecutive days of 15, 1.5 min episodes at 9% O2 (AIH) alternating with 21% O2 at 1 min intervals
  Arms: Repetitive Acute Intermittent Hypoxia
Other: SHAM Acute Intermittent Hypoxia — 5 consecutive days of 15, 1.5 min episodes at 21% O2 (SHAM AIH) alternating with 21% O2 at 1 min intervals
  Arms: SHAM Acute Intermittent Hypoxia

SUMMARY:
The goal of this study is to examine the effect of repetitive acute intermittent hypoxia on motor learning abilities in able-bodied individuals for subsequent study in individuals with incomplete spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old (the latter to reduce likelihood of heart disease);
* Medically stable with medical clearance from physician to participate;
* Motor-incomplete spinal cord injuries at or below C2 and at or above L5;
* AIS A-D at initial screen, or other non-traumatic spinal cord injury disorders (e.g. multiple sclerosis, ALS, tumors, acute transverse myelitis, etc.);
* More than 1 year since iSCI to minimize confounds of spontaneous neurological recovery;
* Ability to advance one step overground with or without assistive devices;

Exclusion Criteria:

* Severe concurrent illness or pain;
* Recurrent autonomic dysreflexia;
* History of cardiovascular/pulmonary complications;
* Concurrent physical therapy;
* Pregnant at time of enrollment or planning to become pregnant;
* Untreated painful musculoskeletal dysfunction, fracture or pressure sore;
* History of seizures or epilepsy;
* Recurring headaches;
* Concussion within the last six months;
* Depression or manic disorders
* Metal implants in the head, or pacemaker.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado, Boulder, Colorado

REFERENCES:
- [Result] Bogard AT, Hembree TG, Pollet AK, Smith AC, Ryder SC, Marzloff GE, Tan AQ. Intermittent hypoxia-induced enhancements in corticospinal excitability predict gains in motor learning and metabolic efficiency. Sci Rep. 2025 Feb 24;15(1):6614. doi: 10.1038/s41598-025-90890-8. PMID 39994358
- [Result] Bogard AT, Hemmerle MR, Smith AC, Tan AQ. Enhanced motor learning and motor savings after acute intermittent hypoxia are associated with a reduction in metabolic cost. J Physiol. 2024 Nov;602(21):5879-5899. doi: 10.1113/JP285425. Epub 2023 Nov 20. PMID 37983629
- See also: Related Info — https://doi.org/10.1038/s41598-025-90890-8

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited through advertisements in Colorado, with recruitment occurring from May 2022 through January 2025. A total of 56 participants were enrolled across both studies. Part 1: Motor Learning (N = 30) & Part 2: Corticospinal Indices of Motor Learning (N = 26).
Pre-assignment Details: Participants were randomly assigned to their respective groups and completed either AIH, SHAM, or no treatment before undergoing motor learning assessments using a split-belt treadmill paradigm. Qualifying participants also received corticospinal excitability assessments using transcranial magnetic stimulation (TMS).
Groups:
- Control Group: No AIH or SHAM exposure
Period: Overall Study
Arm/Group | Repetitive Acute Intermittent Hypoxia | SHAM Acute Intermittent Hypoxia | Control Group
Started | 28 | 13 | 15
Completed | 28 | 13 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Repetitive Acute Intermittent Hypoxia | SHAM Acute Intermittent Hypoxia | Control Group | Total
Number analyzed (Participants) | 28 | 13 | 15 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 2 | 3
  Between 18 and 65 years | 28 | 12 | 13 | 53
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 6 | 8 | 30
  Male | 12 | 7 | 7 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 26 | 12 | 13 | 51
  More than one race | 2 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Corticospinal Excitability
Description: Transcranial magnetic stimulation (TMS) can be applied over the primary motor cortex to examine changes in corticospinal excitability. The downstream muscle activation can be recorded with surface EMG as a motor-evoked potential (MEP). The peak-to-peak MEP amplitude (mV) is as an index of corticospinal excitability.
  A randomized sequence of TMS intensities can be applied over the primary motor cortex, ranging from 90-140% of the participants' resting motor threshold (RMT). The mean MEP amplitude will be plotted against the corresponding stimulation intensity to produce the recruitment curve. The area under the recruitment curve is an additional index of corticospinal excitability (mV/% RMT).
Time Frame: We will measure TMS before the start of 5 consecutive days of AIH or SHAM treatment. We will measure TMS within 24 hours of the final treatment.
Population: A total of 56 participants were enrolled for this study: Part 1: Motor Learning (N = 30; AIH group + control group) & Part 2: Corticospinal Indices of Motor Learning (N = 36; AIH group + SHAM group). Changes in corticospinal excitability reflect the results from Part 2 of the study, which consisted of an AIH group and a SHAM group (i.e., blinded normoxia).
Measure: Mean (Standard Error); unit: mV*percentage of RMT
Arm/Group | Repetitive Acute Intermittent Hypoxia | SHAM Acute Intermittent Hypoxia
Number analyzed (Participants) | 13 | 13
mV*percentage of RMT | 0.528 (0.188) | 0.132 (0.188)
Statistical Analysis 1: Comparison: Repetitive Acute Intermittent Hypoxia vs SHAM Acute Intermittent Hypoxia; Test type: Superiority; p = 0.0098, Mixed Models Analysis; Mean Difference (Net) = 0.528, Standard Error of Mean 0.188
Statistical Analysis 2: Comparison: Repetitive Acute Intermittent Hypoxia; Linear regression analyses performed with the change in the MEP amplitude versus step length asymmetry; Test type: Other; p = 0.014, Regression, Linear; Adjusted R-squared = 0.418
Statistical Analysis 3: Comparison: Repetitive Acute Intermittent Hypoxia; Linear regression analyses performed with the change in the MEP amplitude versus step time asymmetry; Test type: Other; p = 0.006, Regression, Linear; Adjusted R-squared = 0.496
Statistical Analysis 4: Comparison: Repetitive Acute Intermittent Hypoxia; Linear regression analyses performed with the change in the MEP amplitude versus changes in net metabolic power; Test type: Other; p = 0.001, Regression, Linear; Adjusted R-squared = 0.666

2. Primary Outcome: Step Length Asymmetry
Description: Step length asymmetry will be quantified as the ratio of the normalized difference in step lengths between the fast and slow legs during split-belt motor adaptation: (Fast leg - Slow leg step length) / (Fast leg + Slow leg step length).
Time Frame: We will compare asymmetry 15 minutes after the final AIH treatment to asymmetry following no treatment (control group).
Population: A total of 56 participants were enrolled for this study: Part 1: Motor Learning (N = 30; AIH group + control group) & Part 2: Corticospinal Indices of Motor Learning (N = 36; AIH group + SHAM group). Changes in step length asymmetry reflect the results from Part 1 of the study, which consisted of an AIH group and a control group.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Repetitive Acute Intermittent Hypoxia | Control Group
Number analyzed (Participants) | 15 | 15
Ratio | -0.052 (0.023) | -0.0478 (0.024)
Statistical Analysis 1: Comparison: Repetitive Acute Intermittent Hypoxia vs Control Group; Test type: Superiority; p = 0.744, ANOVA; Median Difference (Net) = -0.0042, Standard Deviation 0.0232

3. Primary Outcome: Step Time Asymmetry
Description: Step time asymmetry will be quantified as the ratio of the normalized difference in step times between the fast and slow legs during split-belt motor adaptation: (Fast leg - Slow leg step time) / (Fast leg + Slow leg step time).
Time Frame: We will compare asymmetry 15 minutes after the final AIH treatment to asymmetry following no treatment (control group).
Population: A total of 56 participants were enrolled for this study: Part 1: Motor Learning (N = 30; AIH group + control group) & Part 2: Corticospinal Indices of Motor Learning (N = 36; AIH group + SHAM group). Changes in step time asymmetry reflect the results from Part 1 of the study, which consisted of an AIH group and a control group.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Repetitive Acute Intermittent Hypoxia | Control Group
Number analyzed (Participants) | 15 | 15
Ratio | 0.0781 (0.021) | 0.0681 (0.0252)
Statistical Analysis 1: Comparison: Repetitive Acute Intermittent Hypoxia vs Control Group; Test type: Superiority; p = 0.269, ANOVA; Mean Difference (Net) = 0.01, Standard Deviation 0.0231

4. Primary Outcome: Net Metabolic Power
Description: Using expired gas analyses, we will calculate net metabolic power by inputting steady-state values for V̇O₂ and V̇CO₂ into standard regression equations (W), subtracting resting values, and normalizing the result to each participant's body weight (kg).
Time Frame: We will compare net metabolic power 15 minutes after the final AIH treatment to asymmetry following no treatment (control group).
Population: A total of 56 participants were enrolled for this study: Part 1: Motor Learning (N = 30; AIH group + control group) & Part 2: Corticospinal Indices of Motor Learning (N = 36; AIH group + SHAM group). Changes in net metabolic power reflect the results from Part 1 of the study, which consisted of an AIH group and a control group.
  One participant was excluded from metabolic analysis due to RER > 1.0, violating assumption that primarily oxidative pathways were being utilized.
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | Repetitive Acute Intermittent Hypoxia | Control Group
Number analyzed (Participants) | 15 | 15
W/kg | 3.87 (0.397) | 4.27 (0.766)
Statistical Analysis 1: Comparison: Repetitive Acute Intermittent Hypoxia vs Control Group; Test type: Superiority; p = 0.020, ANOVA; Median Difference (Net) = -0.4, Standard Deviation 0.681

ADVERSE EVENTS:
Time Frame: 2 years 6 months
Description: No serious adverse events were encountered during clinical trial period (see table). Strict inclusion and exclusion criteria were adhered such that intervention does not increase of All-Cause Mortality. Study does not increase risk of adverse events as a consequence of participation.
Groups:
- SHAM Acute Intermittent Hypoxia: Blinded normoxia (5 consecutive days of 21% O2)
Arm/Group | Repetitive Acute Intermittent Hypoxia | Control Group | SHAM Acute Intermittent Hypoxia
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/28 | 0/15 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT05341466/Prot_SAP_000.pdf